CLINICAL TRIAL: NCT01694407
Title: A Phase I Clinical Trial Assessing the Safety, Pharmacokinetics, Pharmacodynamics, and Disintegration Time of Vaginal Tablets Containing Tenofovir and/or Emtricitabine
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics, and Disintegration Time of Vaginal Tablets Containing Tenofovir and/or Emtricitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A11-117
Record Dates: First submitted 2012-07-17; First posted 2012-09-27 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: HIV
Keywords: Prevention
MeSH Terms: interventions — Tenofovir; Emtricitabine; Racivir

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TFV Alone Vaginal Tablet (Active Comparator)
  Interventions: Drug: Tenofovir (TFV) Alone Vaginal Tablet
- Emtricitabine (FTC) Alone Vaginal Tablet (Active Comparator)
  Interventions: Drug: Emtricitabine (FTC) Alone Vaginal Tablet
- TFV Combined with FTC Vaginal Tablet (Active Comparator)
  Interventions: Drug: TFV and FTC Combined Vaginal Tablet
- Placebo Vaginal Tablet (Placebo Comparator)
  Interventions: Drug: Placebo Vaginal Tablet

INTERVENTIONS:
Drug: Tenofovir (TFV) Alone Vaginal Tablet — vaginal tablet containing 40 mg of TFV
  Arms: TFV Alone Vaginal Tablet
Drug: Emtricitabine (FTC) Alone Vaginal Tablet — Vaginal Tablet containing 40 mg of TFV
  Arms: Emtricitabine (FTC) Alone Vaginal Tablet
Drug: TFV and FTC Combined Vaginal Tablet — vaginal tablet with 40 mg TFV and 40 mg FTC
  Arms: TFV Combined with FTC Vaginal Tablet
Drug: Placebo Vaginal Tablet — Vaginal Tablet containing no drug
  Arms: Placebo Vaginal Tablet

SUMMARY:
This prospective, double-blinded, randomized, parallel cohort study will examine the genital and systemic safety, pharmacokinetics (PK), pharmacodynamics (PD), disintegration and disappearance times, and acceptability of four vaginal tablets: 1) Tenofovir (TFV) alone; 2) Emtricitabine (FTC) alone; 3) TFV combined with FTC; and 4) placebo. Participants will be randomized to treatment group, to number of tablets to be inserted in the Single Use Phase (1 tablet or 1 tablet followed by a second tablet two hours later to mimic the BAT24 dosing regimen), and to one of four collection time points (2, 4, 6, or 24 hours after tablet insertion) for assessments only after the last dose of the Multiple Use Phase.

In the Single Use Phase of the study, the participant will insert one tablet in the clinic to estimate times to disintegration and disappearance. Those randomized to two tablets will insert a second tablet 2 hours later. In all women, sample collection will occur 5 hours after the initial tablet insertion.

In the Multiple Use Phase of the study, participants will insert a tablet once daily for 14 days. The 1st, 7th, and 14th tablets will be inserted in the clinic; the remaining tablets will be inserted at home. The clinic will call the participant on day 3 of the multiple use phase to ask about any symptoms the participant may be experiencing. Each insertion in the clinic will be followed by sample collection and, at Visits 4 and 6, colposcopy at the participant's assigned time point.

DETAILED DESCRIPTION:
Objectives:

Primary:

* To assess genital safety after a single use (consisting of one tablet in half of participants and one tablet followed by a second tablet two hours later in the other half) and during and after two weeks of daily tablet use
* To assess systemic safety after two weeks of daily tablet use
* To assess the pharmacokinetics (PK) of TFV and FTC after a single use (as defined above) and during and after two weeks of daily tablet use

Secondary:

* To estimate the time needed for tablet disintegration and the time needed for full tablet disappearance
* To assess acceptability of the tablet
* To assess indicators of the pharmacodynamics (PD) of TFV and FTC in vitro using biological samples (fluids) from study participants obtained before use, after a single (use as define above), and after two weeks of daily tablet use

Exploratory:

•To assess exploratory indicators of the PD of TFV and FTC in vitro using biological samples (tissues) from study participants obtained before use, after a single use (as defined above), and after two weeks of daily tablet use

ELIGIBILITY:
Inclusion Criteria:

* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes)
* Currently having regular menstrual cycles of 25 - 35 days by participant report
* History of Pap smears and follow-up consistent with American Congress of Obstetricians and Gynecologist (ACOG) practice guidelines #99 and #109 or willing to undergo a Pap smear at Visit 1
* Protected from pregnancy, meaning one of the following:

  * Sexually abstinent and planning to remain abstinent for the duration of the study;
  * In a monogamous heterosexual relationship for at least four months with a partner who is not known to be HIV positive and has no known risks for sexually transmitted infections (STIs) and:
* Couple is using condoms and is willing to use non-spermicidally lubricated condoms throughout the study or
* One partner is sterilized; or

  * In a monogamous same sex relationship for at least four months with a partner who is not known to be HIV positive and has no known risks for STIs.
* Willing to abstain from vaginal activity as follows:

Starting 48 hours before Visit 2 until the sixth day after Visit 2 Starting 48 hours before Visit 3 until the sixth day after Visit 3 Starting 48 hours before Visit 4 until the sixth day after Visit 6

* Willing to abstain from the use of any vaginal product other than the study product including spermicides, lubricants, and douches starting 48 hours before Visit 2 until the sixth day after Visit 6 (tampons may be used, but for menses only)
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy colposcopy and genital tract sample collection
* Negative urine pregnancy test
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

* History of hysterectomy
* Currently pregnant or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome
* Use of any hormonal contraceptive method in the last 30 days (oral, transdermal, transvaginal, implant, or hormonal intrauterine contraceptive device)
* Injection of Depo-Provera in the last 6 months
* Current use of IUD
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the study products, topical anesthetic, or allergy to both silver nitrate and Monsel's solution
* In the last six months, diagnosed with or treated for any STI or pelvic inflammatory disease. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility
* Nugent score greater than or equal to 7 at Visit 1 or symptomatic bacterial vaginosis (BV) as defined by Amsel's criteria at Visit 1 or 2
* Symptomatic vulvovaginal candidiasis or symptomatic urinary tract infection (UTI)
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea or Chlamydia trachomatis
* Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for an STI
* Positive test for HIV
* Positive test for Hepatitis B surface antigen (HBsAg)
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.)
* Known current drug or alcohol abuse which could impact study compliance
* Grade 1 or higher laboratory abnormality, per the August 2009 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events (AEs)
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, antifungals, antivirals (e.g., acyclovir or valacyclovir) or antiretrovirals (e.g., Viread, Atripla, Emtriva, Complera). Note: Participants should avoid non-steroidal anti-inflammatory drugs (NSAIDs) except for treatment of dysmenorrhea during menses. Participants may use Tylenol® on an as-needed but not daily basis during the study.
* Participation in any other investigational trial (device, drug, or vaginal trial) within the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
* Abnormal finding on laboratory or physical examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in Genitourinary AEs | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Genitourinary AEs, moderate to severe
Changes on physical examination and colposcopy | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Changes on physical examination and colposcopy
Changes Soluble markers of mucosal immunity, immune cell numbers, & characteristics in CVL | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Changes Soluble markers of mucosal immunity, immune cell numbers, & characteristics in CVL
Changes in Number, phenotype and activation status of immune cells in cervicovaginal mucosa | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Changes in Number, phenotype and activation status of immune cells in cervicovaginal mucosa
Changes in Mucosal histology in cervicovaginal tissue | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Changes in Mucosal histology in cervicovaginal tissue
Changes in Changes in microflora | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Changes in Changes in microflora (semiquantitative cultures and unculturable species)
Changes in Systemic laboratory tests | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Changes in Systemic laboratory tests
TFV & FTC concentrations in plasma, vaginal aspirate, & genital tissue | 5 hours after first tablet insertion
  TFV & FTC concentrations in plasma, vaginal aspirate, & genital tissue Pharmacokinetics Mean (SD) and Median (Min, Max, C-Max, T-Max) of TFV and FTC in blood, vaginal aspirate,and genital tissue at Visit 2, 3, 4, 5, 6
TFV-DP and FTC-TP concentrations in PBMCs, endocervical cells, & genital tissue | 5 hours after first tablet insertion
  TFV-DP and FTC-TP concentrations in PBMCs, endocervical cells, & genital tissue Pharmacokinetics C-Max and T-Max of Blood TFV and FTC levels at single dose phase, by site and overall, Evaluable Population
TFV & FTC concentrations in plasma, vaginal aspirate, & genital tissue | after 7th daily tablet
  TFV & FTC concentrations in plasma, vaginal aspirate, & genital tissue Pharmacokinetics Mean (SD) and Median (Min, Max, C-Max, T-Max) of TFV and FTC in blood, vaginal aspirate,and genital tissue at Visit 2, 3, 4, 5, 6
TFV & FTC concentrations in plasma, vaginal aspirate, & genital tissue | after 14 daily tablet insertion
  TFV & FTC concentrations in plasma, vaginal aspirate, & genital tissue Pharmacokinetics Mean (SD) and Median (Min, Max, C-Max, T-Max) of TFV and FTC in blood, vaginal aspirate,and genital tissue at Visit 2, 3, 4, 5, 6
TFV-DP and FTC-TP concentrations in PBMCs, endocervical cells, & genital tissue | after 7th daily tablet
  TFV-DP and FTC-TP concentrations in PBMCs, endocervical cells, & genital tissue Pharmacokinetics C-Max and T-Max of Blood TFV and FTC levels at single dose phase, by site and overall, Evaluable Population
TFV-DP and FTC-TP concentrations in PBMCs, endocervical cells, & genital tissue | after 14th daily tablet
  TFV-DP and FTC-TP concentrations in PBMCs, endocervical cells, & genital tissue Pharmacokinetics C-Max and T-Max of Blood TFV and FTC levels at single dose phase, by site and overall, Evaluable Population

SECONDARY OUTCOMES:
Pharmacodynamics | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Anti-HIV and anti-HSV activity in CVL
  Anti-HIV and anti-HSV activity as a percent of anti-HIV and anti-HSV activity before exposure to test product
Disintegration | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Medians and interquartile ranges of (a) time to disintegration (tablet no longer coherent but residual product is visible) and (b) time to complete disappearance
Acceptability | 5 hours after first tablet insertion and after 7th and 14th daily tablet
  Responses on acceptability questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, Study Director — CONRAD
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Clinical Research Center, Eastern Virginia Medical School, Norfolk, Virginia